CLINICAL TRIAL: NCT02923817
Title: Phase I-II Clinical Trial Using Bone Marrow-derived Mononuclear Cells for Spinal Cord Injury
Brief Title: Clinical Trial Using Bone Marrow-derived Mononuclear Cells for Spinal Cord Injury
Acronym: DNH
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Da Nang Hospital (Other)
Collaborators: Kitano Hospital (Unknown); Translational Research Center for Medical Innovation, Kobe, Hyogo, Japan (Other)
Responsible Party: Principal Investigator, Ngoc Ba Nguyen, Vice-director, Da Nang Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DNHSCI124HP
Record Dates: First submitted 2016-10-03; First posted 2016-10-05 (Estimated); Last update posted 2017-01-10 (Estimated); Status verified 2017-01

CONDITIONS: Spinal Cord Injuries
Keywords: spinal cord injury; autologous transplants; bone marrow derived mononuclear cells
MeSH Terms: conditions — Spinal Cord Injuries

ARMS (1):
- Treatment (Experimental)
  Interventions: Biological: Transplantation of autologous bone marrow-derived mononuclear cells by lumbar injection

INTERVENTIONS:
Biological: Transplantation of autologous bone marrow-derived mononuclear cells by lumbar injection

SUMMARY:
The purpose of study is to determine whether autologous mononuclear cells deriving from the bone marrow are effective in the treatment of spinal cord injury.

DETAILED DESCRIPTION:
Recruitment process:

The investigators selects the candidate of the study that fulfill the inclusion criteria and not violate any exclusion criteria from patients with spinal cord injury that admitted to the department of neurosurgery - Danang hospital. The investigators then ask the patients and patients family for informed consent. The patients that submit the informed consent to participate is recruited to the study.

Procedure description:

The patients is moved to operation theater at the day of the procedure. The bone marrow of the patients is harvested by two investigators. The mononuclear cells of the bone marrow is extracted from the bone marrow by using gravity centrifugation with Ficoll Paque 1.073. The mononuclear cells is transferred to 5 mL syringe and handed back to the investigator. The investigator will transplant the whole cell preparation back to the patients by lumbar injection.

A final supernatant layer of the preparation is also sent to the lab for microbiological and endotoxin testings. One small portion of the cell preparation is sent to the laboratory for cell count and cluster of distribution tests.

The patient is transferred back to the patient room and monitor for the outcomes at 2 weeks, 4 weeks, 2 months, 4 months, 6 months. All of the data is entered, stored and monitored via the eCB database system of TRI Cente, Kobe.

Data Analysis:

Primary Endpoint:

A list is prepared for each subject with the name of AE developed, its severity and seriousness, causal relationship with the treatment, and outcome. In addition, the incidence of AEs in all cases and the 95% confidence interval are estimated. For each AE type, the incidence, incidence by severity, and incidence by seriousness are calculated in addition to estimation of the rate of each AE and its 95% confidence interval in all cases.

Secondary Endpoint:

Regarding secondary endpoints, the Wilcoxon signed rank test is used to compare the baseline value at registration and value at 6 months after cell transplantation. In addition, assuming the scores in each secondary endpoint to be consecutive scores, a linear mixed model with time point as a fixed effect and cases as random effects is fitted to the data at registration and 2 and 6 months after cell transplantation after assuming an appropriate covariance structure between time points to assess their chronological changes.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with spinal cord injuries classified as A-B on the ASIA impairment scale
2. Patients injured 3 weeks to 1 year previously
3. Patients with partial spinal cord injury demonstrated by diagnostic imaging
4. Patients aged between 20 and 60 years at the acquisition of informed consent
5. Patients who submitted written informed consent by themselves

Exclusion Criteria:

1. Patients with a completely transected spinal cord
2. Patients with central spinal cord injury
3. Patients with organ failure with SOFA score of 3 points or higher
4. Patients in whom hepatitis B, hepatitis C, human immunodeficiency virus infection, or leukemia infection cannot be denied
5. Patients with malignant tumour or a history of malignant tumour within 5 years
6. Patients with following disease/disorder:

   Myeloproliferative disorder or myelodysplastic syndrome Poorly controlled ischemic heart disease Autoimmune disease Spinal stenosis Limb paralysis due to central nervous system disorder not attributed to spinal cord injury Hepatic dysfunction Renal dysfunction Poorly controlled psychiatric disorder Complex multiple trauma
7. Patients who are participating in other clinical trials or who completed participation within 6 months
8. Patients who are pregnant or possibly pregnant
9. Other patients who are judged to be ineligible by investigators

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-09; Primary Completion 2018-12 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Safety profile and adverse effects of the procedure | 6 months from the time when patients receive the treatment
  Causal relationship, incidence, severity, and seriousness of all adverse events (AEs) experienced following cell transplantation up to the day of the final observation are assessed.

SECONDARY OUTCOMES:
Motor function | At 2 weeks, 4 weeks, 2 months, 4 months, 6 months after the transplantation
  Motor function score in the neurological classification of spinal cord injury: Amount of change from the time of registration to 6 months after cell transplantation
Sensory function | At 2 weeks, 4 weeks, 2 months, 4 months, 6 months after the transplantation
  Sensory function score in the neurological classification of spinal cord injury (light touch sensation score + pinprick sensation score): Amount of change from the time of registration to 6 months after cell transplantation
ASIA Impairment Scale | At 2 weeks, 4 weeks, 2 months, 4 months, 6 months after the transplantation
  Change on the ASIA impairment scale from the time of registration to 6 months after cell transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Ba Ngoc Nguyen, MD, Principal Investigator — Danang Hospital; Yoshihisa Suzuki, MD, PhD., Study Director — Kitano Hospital
Locations (1):
- Danang Hospital, Da Nang, Da Nang City, Vietnam